CLINICAL TRIAL: NCT02573532
Title: Basel Incidence, Patient Characteristics, Outcome and Possible Strategies to Improve Outcome of Perioperative Myocardial Injury After Non-cardiac Surgery: 1-Year Follow-up
Brief Title: Incidence and Outcome of Perioperative Myocardial Injury After Non-cardiac Surgery
Acronym: BASEL-PMI
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Cantonal Hospital of Aarau, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: BASEL-PMI
Record Dates: First submitted 2015-10-01; First posted 2015-10-09 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Perioperative Myocardial Injury
Keywords: myocardial ischemia/diagnosis; myocardial ischemia/epidemiology; perioperative; perioperative complications/diagnosis; prognosis
MeSH Terms: conditions — Myocardial Ischemia; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study includes patients undergoing major non-cardiac surgery, and screens them for the occurrence of perioperative myocardial injuries (PMI). Incidence, patient characteristics, pathophysiology, potential prevention and therapy strategies and 1-year outcomes of PMI will be described.

DETAILED DESCRIPTION:
Background: Worldwide more than 230 million surgical operations are performed each year. Despite advances in all fields of medicine, there is still a significant risk of death related to major non-cardiac surgical procedures. The observed 30-day mortality depends on patient- as well as procedural factors and ranges between 1% and 10%. Cardiovascular complications, particularly perioperative myocardial injury/infarction (PMI) seem to be major contributors to about a third of all deaths. PMI may differ from spontaneous acute myocardial infarction (AMI). The vast majority of patients experiencing PMI do NOT have acute chest pain or other symptoms typical for AMI likely because they are narcotized or sedated and random ECGs are often not informative. Accordingly, most patients with PMI are currently not detected in routine clinical practice. Missed diagnosis is invariably associated with missed opportunity for the initiation of treatment. As most patients with PMI are missed in routine clinical care, the true incidence of and outcome after PMI are largely unknown. Prior studies have often not obtained a baseline sample and thus have suggested that all cTn elevations are likely due to AMI which may exaggerate the numbers. In addition, usually conventional less sensitive assays have been used. Further, the predominant pathophysiology of PMI is currently unknown. It has been suggested that type II MI characterized by coronary perfusion pressure mismatch and not type I MI characterized by acute thrombotic coronary occlusion is the predominate mechanism. However, autopsy data suggest that plaque rupture is more common. Thus, it may be that type 2 AMI is more common but that the modest incidence of type 1 AMI is not dangerous prognostically.

Aim: To explore the incidence, patient characteristics, pathophysiology, potential prevention and therapy strategies and long-term outcome of PMI after major non-cardiac surgery

Methodology: Consecutive high-risk patients undergoing major non-cardiac surgery will be included and followed for one year for the occurrence of all-cause death and other major adverse cardiac events. Patients receive a standardized assessment of cardiovascular status and systematic perioperative screening for PMI using high sensitivity cardiac troponin T (hs-cTnT) at baseline prior to surgery, as well as on day 1 and day 2 after surgery. Acute cardiac injury will be defined as an absolute increase in h/s-cTn of the 99th percentile of healthy individuals for the respective assay above baseline cTn-value or between two postoperative values if the preoperative value is missing. A search for possible alternative causes for hs-cTnT elevations will be aggressively sought if a rising pattern of values is detected. Two independent experts will adjudicate the most likely cause of PMI using all clinical information pertaining to the individual patient including the 12-lead ECG, peak hs-cTnT blood concentrations, coronary angiography and myocardial perfusion scanning. Influence of PMI on occurrence of all-cause death will be assessed using multivariate Cox-proportional hazards analysis. Further, pre-operative and post-operative prediction models for death, major adverse cardiac events, and PMI shall be derived using a derivation-validation design.

Potential Significance: This study will generate scientific data that have major scientific implications by contributing to closing current knowledge gaps concerning the influence of PMI on long-term mortality as well as the incidence, patient characteristics, and pathophysiology of PMI after non-cardiac surgery. This knowledge will have immediate clinical implications as it could e.g. lead to major changes in perioperative management with reconsiderations of the necessary target blood pressure to avoid coronary perfusion mismatch and consecutive cardiac injury.

ELIGIBILITY:
Inclusion criteria

* Patients received a perioperative hs-cTnT screening for PMI
* Patient consent available Exclusion criteria
* Patient's refusal

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients that underwent a systematic approach to PMI detection at the participating hospitals as clinical routine will be included.
  The screening consists of a pre-operative "baseline" measurement of hs-cTnT within 30 days prior to surgery, and two post-operative measurements taken on the first and second day after surgery. Screening is done in patients requiring hospitalization >24 hours after surgery AND (aged ≥ 65 years OR history of coronary artery disease OR peripheral artery occlusive disease OR cerebrovascular disease). Patients are seen by a cardiologist in case of detection of a PMI.
Sampling Method: Probability Sample
Enrollment: 19645 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Deaths in one year after non-cardiac surgery in patients with and without PMI | 1 year

SECONDARY OUTCOMES:
MACE in one year after non-cardiac surgery in patients with and without PMI | 1 year
  MACE is defined as a composite of death, acute myocardial infarction, life-threatening arrhythmia (cardiac arrest, sustained ventricular tachycardia, atrioventricular (AV) -block III), or acute heart failure (requiring admission to a hospital or intra-hospital transfer to the intensive care unit) within one year. Two independent cardiologists or anaesthesiologists will adjudicate all MACE.
Incidence of PMI within a screening program in high-risk patients undergoing major non-cardiac surgery | 3 days after surgery
  PMI is defined as an absolute increase in h/s-cTn of the 99th percentile of healthy individuals for the respective assay above baseline cTn-value or between two postoperative values if the preoperative value was missing. PMI will be further classified as type I myocardial infarction, type II myocardial infarction, or myocardial injury due to non-cardiac causes.
Number of patients with PMI with ischemic symptoms and signs detected in a screening program in high-risk patients undergoing major non-cardiac surgery | 3 days after surgery
  Patients with PMI are evaluated for: presence of chest pain, atypical symptoms, palpitations, dyspnea, edema, or nausea; ST-changes, Q-waves, T-wave abnormalities, new bundle branch block
Number of patients with PMI with management changes after screening-induced consultation | 3 days after surgery, followed for 1 year
  Changes in management can be: changes in medication, intensification of surveillance, call for use of coronary angiography, myocardial stress testing, other, or none
Generate a pre- and an immediate postoperative prediction score for occurrence of major adverse cardiac events including PMI | 1 year
Costs related to the introduction of perioperative hs-cTnT screening. | 1 year
  Health system costs of implementation of screening is calculated as number of interventions initiated additionally to routine care after screening
Derive and validate a risk score in patients with different subtypes of PMI for the occurrence of major cardiac adverse events to inform treatment decisions. | 1 year
  Endpoint: percentage of correctly classified patients in validation cohort.
Derive and validate an improved diagnostic screening approach for detection of PMI. | 3 days after surgery
  Endpoint: sensitivity and specificity for PMI.
Evaluate the effect of pre-operative medication use. | 3 days after surgery
  Endpoint: number of patients undergoing elective non-cardiac surgery suffering PMI (cardiac origin) after non-cardiac surgery with vs without pre-operative statin/RAAS blocker/β-blocker therapy.
Evaluate the effect of post-PMI medication on outcome of PMI. | 1 year
  Endpoint: death and MACE in patients suffering PMI (cardiac origin) with vs without statin/RAAS blocker/β-blocker therapy.
Description of PMI subtypes and potential diagnostic criteria available at time of PMI detection. | 3 days after surgery
Validate the diagnosis of PMI within a screening program in high-risk patients undergoing major non-cardiac sur-gery with other troponin assays. | 3 days after surgery
  PMI is defined as an absolute increase in h/s-cTn of the 99th percentile of healthy individuals for the respective assay above baseline cTn-value or between two postoperative values if the preoperative value was missing.

OTHER OUTCOMES:
Estimate potential effect of detection and management of PMI on major adverse cardiac events by a screening program implemented within clinical routine | 1 year
Compare cardiac troponin T and I in the detection of PMI | 3 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christian Müller, MD, Prof, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Champetier A, Lopez-Ayala P, Puelacher C, Durak K, Kaplan E, Gualandro D, Glarner N, Pargger M, Hure G, Burri-Winkler K, Bolliger D, Steiner LA, Scharen S, Mujagic E, Clauss M, Mueller AM, Lardinois D, Boeddinghaus J, Mahfoud F, Strebel I, Mueller C. External validation of PreOpNet to predict 30-day mortality after major non-cardiac surgery using digital electrocardiogram. NPJ Digit Med. 2025 Oct 16;8(1):613. doi: 10.1038/s41746-025-01983-7. PMID 41102258
- [Derived] Durak K, Burri-Winkler K, Hure G, Strebel I, Reinhardt J, Thommen V, Pargger M, Glarner N, Haziri F, Seeberger E, Doyle N, Bolliger D, Steiner LA, Mujagic E, Lardinois D, Scharen S, Mueller A, Mahfoud F, Gualandro DM, Puelacher C, Mueller C. Robotic process automation to identify patients at high risk for perioperative myocardial infarction or injury: a prospective, blinded, paired reader-controlled single-centre study. Br J Anaesth. 2025 Nov;135(5):1153-1160. doi: 10.1016/j.bja.2025.07.035. Epub 2025 Jul 31. PMID 40750466
- [Derived] Glarner N, Puelacher C, Gualandro DM, Pargger M, Hure G, Maiorano S, Strebel I, Fried S, Bolliger D, Steiner LA, Lampart A, Lurati Buse G, Mujagic E, Lardinois D, Kindler C, Guerke L, Schaeren S, Mueller A, Clauss M, Buser A, Hammerer-Lercher A, Mueller C; Basel-PMI Investigators. Association of preoperative beta-blocker use and cardiac complications after major noncardiac surgery: a prospective cohort study. Br J Anaesth. 2024 Jun;132(6):1194-1203. doi: 10.1016/j.bja.2024.02.023. Epub 2024 Apr 15. PMID 38627137
- [Derived] Glarner N, Puelacher C, Gualandro DM, Lurati Buse G, Hidvegi R, Bolliger D, Lampart A, Burri K, Pargger M, Gerhard H, Weder S, Maiorano S, Meister R, Tschan C, Osswald S, Steiner LA, Guerke L, Kappos EA, Clauss M, Filipovic M, Arenja N, Mueller C; for the BASEL-PMI Investigators. Guideline adherence to statin therapy and association with short-term and long-term cardiac complications following noncardiac surgery: A cohort study. Eur J Anaesthesiol. 2023 Nov 1;40(11):854-864. doi: 10.1097/EJA.0000000000001903. Epub 2023 Sep 25. PMID 37747427
- [Derived] Puelacher C, Gualandro DM, Glarner N, Lurati Buse G, Lampart A, Bolliger D, Steiner LA, Grossenbacher M, Burri-Winkler K, Gerhard H, Kappos EA, Clerc O, Biner L, Zivzivadze Z, Kindler C, Hammerer-Lercher A, Filipovic M, Clauss M, Gurke L, Wolff T, Mujagic E, Bilici M, Cardozo FA, Osswald S, Caramelli B, Mueller C; BASEL-PMI Investigators. Long-term outcomes of perioperative myocardial infarction/injury after non-cardiac surgery. Eur Heart J. 2023 May 14;44(19):1690-1701. doi: 10.1093/eurheartj/ehac798. PMID 36705050
- [Derived] Arslani K, Gualandro DM, Puelacher C, Lurati Buse G, Lampart A, Bolliger D, Schulthess D, Glarner N, Hidvegi R, Kindler C, Blum S, Cardozo FAM, Caramelli B, Gurke L, Wolff T, Mujagic E, Schaeren S, Rikli D, Campos CA, Fahrni G, Kaufmann BA, Haaf P, Zellweger MJ, Kaiser C, Osswald S, Steiner LA, Mueller C; BASEL-PMI Investigators. Cardiovascular imaging following perioperative myocardial infarction/injury. Sci Rep. 2022 Mar 15;12(1):4447. doi: 10.1038/s41598-022-08261-6. PMID 35292719
- [Derived] Lurati Buse GAL, Puelacher C, Gualandro DM, Kilinc D, Glarner N, Hidvegi R, Bolliger D, Arslani K, Lampart A, Steiner LA, Kindler C, Wolff T, Mujagic E, Guerke L, Mueller C; Incidence and Outcome of Perioperative Myocardial Injury After Non-cardiac Surgery (BASEL-PMI) Investigators. Adherence to the European Society of Cardiology/European Society of Anaesthesiology recommendations on preoperative cardiac testing and association with positive results and cardiac events: a cohort study. Br J Anaesth. 2021 Sep;127(3):376-385. doi: 10.1016/j.bja.2021.06.027. Epub 2021 Jul 28. PMID 34330416
- [Derived] Sazgary L, Puelacher C, Lurati Buse G, Glarner N, Lampart A, Bolliger D, Steiner L, Gurke L, Wolff T, Mujagic E, Schaeren S, Lardinois D, Espinola J, Kindler C, Hammerer-Lercher A, Strebel I, Wildi K, Hidvegi R, Gueckel J, Hollenstein C, Breidthardt T, Rentsch K, Buser A, Gualandro DM, Mueller C; BASEL-PMI Investigators. Incidence of major adverse cardiac events following non-cardiac surgery. Eur Heart J Acute Cardiovasc Care. 2021 Jun 30;10(5):550-558. doi: 10.1093/ehjacc/zuaa008. Epub 2020 Oct 14. PMID 33620378
- [Derived] Lurati Buse GAL, Puelacher C, Gualandro DM, Genini AS, Hidvegi R, Bolliger D, Arslani K, Steiner LA, Kindler C, Mueller C; BASEL-PMI Investigators. Association between self-reported functional capacity and major adverse cardiac events in patients at elevated risk undergoing noncardiac surgery: a prospective diagnostic cohort study. Br J Anaesth. 2021 Jan;126(1):102-110. doi: 10.1016/j.bja.2020.08.041. Epub 2020 Oct 17. PMID 33081973
- [Derived] Puelacher C, Gualandro DM, Lurati Buse G, Bolliger D, Marbot S, Kindler C, Hammerer-Lercher A, Gurke L, Steiner L, Mueller C. Etiology of Peri-Operative Myocardial Infarction/Injury After Noncardiac Surgery and Associated Outcome. J Am Coll Cardiol. 2020 Oct 20;76(16):1910-1912. doi: 10.1016/j.jacc.2020.08.043. No abstract available. PMID 33059838
- [Derived] du Fay de Lavallaz J, Puelacher C, Lurati Buse G, Bolliger D, Germanier D, Hidvegi R, Walter JE, Twerenbold R, Strebel I, Badertscher P, Sazgary L, Lampart A, Espinola J, Kindler C, Hammerer-Lercher A, Thambipillai S, Guerke L, Rentsch K, Buser A, Gualandro D, Jakob M, Mueller C; BASEL-PMI Investigators. Daytime variation of perioperative myocardial injury in non-cardiac surgery and effect on outcome. Heart. 2019 Jun;105(11):826-833. doi: 10.1136/heartjnl-2018-313876. Epub 2018 Dec 12. PMID 30541757
- [Derived] Puelacher C, Lurati Buse G, Seeberger D, Sazgary L, Marbot S, Lampart A, Espinola J, Kindler C, Hammerer A, Seeberger E, Strebel I, Wildi K, Twerenbold R, du Fay de Lavallaz J, Steiner L, Gurke L, Breidthardt T, Rentsch K, Buser A, Gualandro DM, Osswald S, Mueller C; BASEL-PMI Investigators. Perioperative Myocardial Injury After Noncardiac Surgery: Incidence, Mortality, and Characterization. Circulation. 2018 Mar 20;137(12):1221-1232. doi: 10.1161/CIRCULATIONAHA.117.030114. Epub 2017 Dec 4. PMID 29203498